CLINICAL TRIAL: NCT02022462
Title: A Randomized Controlled Trial of "The Bridge", a Peer Health Navigation Intervention
Brief Title: Project Bridge: Peer Health Navigator Intervention
Acronym: Bridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John Brekke, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bridge2014; PCORI (Other Grant/Funding Number: AD-1304-6650)
Record Dates: First submitted 2013-12-11; First posted 2013-12-27 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Depression; Medical Disorders; Serious Mental Illness
Keywords: Serious mental illnesses; peer navigator; integrated health care
MeSH Terms: conditions — Schizophrenia; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Navigation (Experimental): 151 participants with SMI in the El Camino clinic, operated by Pacific Clinics, were recruited to participate in a 12-month study of Bridge navigation. Participants were randomly assigned to either waitlist control (6 month waitlist with treatment as usual) or immediate intervention with the Bridge. Participants in the immediate treatment group completed three assessments (baseline, 6 months, and 12 months) and, after 6 months, one interview about their health, healthcare, and navigation experiences. Participants in the waitlist control group completed three assessments (baseline, 6 months, 12 months) and one interview about their health, health care, and their experiences using health navigation after 12 months.
  Interventions: Behavioral: Health Navigation
- Waitlist Control (Other): 151 participants with SMI in the El Camino clinic, operated by Pacific Clinics, were recruited to participate in a 12-month study of Bridge navigation. Participants were randomly assigned to either waitlist control (n = 75, 6-month waitlist with treatment as usual then they received the intervention) or immediate intervention with the Bridge (n = 76). Participants in the immediate treatment group completed three assessments (baseline, 6 months, and 12 months) and, after 6 months, one interview about their health, healthcare, and navigation experiences. Participants in the waitlist control group completed three assessments (baseline, 6 months, 12 months) and one interview about their health, health care, and their experiences using health navigation after 12 months.
  Interventions: Behavioral: Health Navigation

INTERVENTIONS:
Behavioral: Health Navigation — Experimental: Immediate peer health navigator intervention vs. waitlist control.
  The immediate peer health navigator intervention group will receive assistance for 6 months and then followed up with after an additional 6 months. Participants will receive training in how to self-manage their physical health and healthcare. The intervention is individualized and the number of contacts by the navigator will be determined by their need level. The waitlist control group will complete a baseline assessment and then wait for 6 months before receiving the peer health navigator intervention. They will complete a follow-up assessment after 6 months of the intervention.

SUMMARY:
The mortality rate among people with Serious Mental Illness (SMI) is 2 to 3 times that of the general population, meaning that those with a serious mental illness die, on average, 25 years earlier than those without an SMI. These deaths are largely attributed to preventable medical conditions, many of which are more common in the SMI population.

The "Bridge" intervention is a peer navigator model that was developed to target factors that negatively impact healthcare access, utilization, and outcomes among individuals with serious mental illness (e.g., severe mood disorders and psychotic disorders). This intervention targets male and female, adult consumers across races/ethnicities and has been utilized by Pacific Clinics (Southern California's largest behavioral healthcare agency) and the Department of Mental Health of Los Angeles County to improve the health and quality of life for their consumers.

Investigators will test the comparative effectiveness of a peer navigator intervention (the Bridge) to treatment as usual. The Bridge navigator intervention is designed to teach SMI consumers the skills to engage health care providers and to overcome motivational deficits in order to improve their health and healthcare use. The specific aims of this application are:

1. To use randomized methods to examine the effectiveness of the Bridge intervention on the health care utilization, satisfaction with care, health status, and health care self-management for a sample of individuals with severe mental illness receiving public mental health services in the community;
2. To use randomized methods to examine the effectiveness of the Bridge intervention on psychological and social well-being for a sample of individuals with severe mental illness receiving public mental health services in the community.

151 participants in an Full Service Partnership (FSP) clinic operated by Pacific Clinics were recruited to participate in an approximately 24-month long study of Bridge navigation. Participants will be randomly assigned to either treatment as usual (waitlist) or immediate intervention with the Bridge.

Participants in both groups will complete three assessments (baseline, 6 months, 12 months) and statistically compared over time. Staff stakeholders (n = 20) will also be interviewed at baseline and every three months of the study in order to ensure that the intervention is being implemented appropriately.

DETAILED DESCRIPTION:
The mortality rate among people with Serious Mental Illness (SMI) is 2 to 3 times that of the general population (DeHert et al., 2011), meaning that those with a serious mental illness die, on average, 25 years earlier than those without a SMI (Parks et al., 2006). There is evidence that these deaths are largely attributed to preventable medical conditions, many of which are more common in the SMI population. System bifurcation, or the separation of mental and physical health services, has been identified as a critical factor that leads to significant health disparities for those with SMI (Bazelon Center for Mental Health Law, 2004).

Grounded in patients' experiences, needs, and voices, investigators seek to generate knowledge about effective interventions, use outcomes that are central to patients and caregivers, attend to issues of implementation and dissemination, and may seek to optimize outcomes in the context of factors such as burden, technology, and stakeholder perspectives. Based on pilot work funded by the UniHealth Foundation, the goal of this Patient Centered Outcomes Research Institute (PCORI) proposal is to test the effectiveness of a peer health navigation intervention (The Bridge) in comparison to usual treatment. The Bridge is a peer-staffed comprehensive healthcare engagement and self management model, situated in an outpatient mental health clinic, where clients are taught the skills to access and manage their healthcare for any condition. The investigators' goal is train clients to successfully engage and navigate the primary health care system as well as other needed health care services (specialty care, lab, and pharmacy). Guided by a version of Gelberg, Andersen, and Leake's (2000) Behavioral Model of Health Service Use for Vulnerable Populations that investigators adapted for the seriously mentally ill (Brekke et al., in press), the Bridge combines three approaches: integrated care, patient education, and cognitive-behavioral skill building with an in vivo (real world) focus.

Investigators conducted a randomized controlled trial comparing 2 groups: a) a treatment as usual waitlist (n =75), and b) the Bridge peer navigator intervention (n=76). Investigators will compare these groups across 3 time points (baseline, 6 months, 1 year) to examine the Bridge's effectiveness at improving health care service use, satisfaction with care, health knowledge, health status, health related self-efficacy, and quality of life. Outcomes will be measured through patient self-report and according to objective measures of health (medical records and insurance claims data).

In addition, investigators conducted interviews every three months with selected stakeholders to assess the degree to which the intervention and the study are succeeding and what challenges have occurred. This will allow for corrections as the study proceeds. Investigators will focus on the factors that will contribute to the implementation and sustainability of the health navigator intervention including: cost, training, supervision, billing issues, and how this position will fit into the organizational model of the clinic. To begin the interview, investigators ask each person interviewed for his or her ideas about what are the critical factors for implementation and sustainability. Finally, investigators conducted exit interviews with each patient as part of their final assessment. Exit interviews focused on the patients' perceptions about the study, how it affected them, what went well, and what challenges they encountered. Each interview should last about 20-30 minutes and was audio-recorded using an encrypted tape recorder. Investigators will use a semi-structured interview guide so that all interviewees are asked the same questions and data are comparable. Basic demographics such as gender, ethnicity, and age will be recorded for all participants.

This PCORI proposal relies on significant stakeholder involvement in the intervention development, project development and management, and in the plans for dissemination and implementation. The ultimate goal is to provide the field a peer-delivered intervention that significantly reduces disparities in the utilization and outcome of health services for the seriously mentally ill and thereby reduce morbidity and mortality in this highly vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Client participants will have diagnoses of serious mental illness and be between the ages of 18-65. All participants must be able to complete assessments in English.
* Staff participants will be between the ages of 18-65 and must be currently employed at Pacific Clinics. All participants must be able to complete assessments in English.
* Medical providers who serve clients of Pacific Clinics will also be interviewed as stakeholders. They will be between the ages of 18-65 and must be employees of a medical provider serving Pacific Clinics' clients.

Exclusion Criteria:

* Clients who are under the age of 18, over the age of 65, who are under conservatorship, cannot give informed consent themselves, or are not receiving mental health services through Pacific Clinics will not be eligible for participation.
* Staff participants must be currently employed at Pacific Clinics and have the capacity to give informed consent themselves.
* Medical providers must be serving Pacific Clinics' clients and have the capacity to give informed consent themselves.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Duris, Study Director — Pacific Clinics Corporate Director, East Valley Division and New Initiatives
Locations (1):
- Pacific Clinics El Camino, Santa Fe Springs, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] Parks J, Svendsen D, Singer P, Foti ME. Morbidity and mortality in people with serious mental illness. Report from the National Association of State Mental Health Program Directors. 2006.
- [Background] Bazelon Center for Mental Health Law. Get it together. How to integrate physical and mental health care for people with serious mental disorders. Washington DC 2004.
- [Background] Gelberg L, Andersen RM, Leake BD. The Behavioral Model for Vulnerable Populations: application to medical care use and outcomes for homeless people. Health Serv Res. 2000 Feb;34(6):1273-302. PMID 10654830

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Navigation: 76 participants with SMI in the El Camino clinic, operated by Pacific Clinics, recruited to participate in a 12 month study of Bridge navigation. Randomly assigned and completed three assessments (baseline, 6 months, and 12 months) and, after 6 months, one interview about their health, healthcare, and navigation experiences.
  Health Navigation: Experimental: Immediate peer health navigator intervention vs. waitlist control.
  The immediate peer health navigator intervention group will receive assistance for 6 months and then followed up with after an additional 6 months. Part
- Waitlist Control: 75 participants with SMI in the El Camino clinic, operated by Pacific Clinics, recruited to participate in a 12-month study of Bridge navigation. Randomly assigned, participants in the waitlist control group completed 3 assessments (baseline, 6 month, 12 months) and one interview about their health, health care, and their experiences using health navigation after 12 months.
Period: Overall Study
Arm/Group | Health Navigation | Waitlist Control
Started | 76 | 75
Completed | 53 | 50
Not Completed | 23 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Navigation | Waitlist Control | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 73 | 149
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.80 (11.30) | 46.47 (10.59) | 45.63 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 46 | 81
  Male | 41 | 29 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 17 | 20 | 37
  Race/Ethnicity: Black | 7 | 5 | 12
  Race/Ethnicity: Hispanic/LatinX | 46 | 44 | 90
  Race/Ethnicity: Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Changed Score on SF-12 Pain Items From Baseline to 6 Months and 12 Months
Description: Changed score on SF-12 pain items from baseline to 6 months and 12 months in active intervention group and changed score from 6 months to 12 months in the waitlist control group. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more pain. A negative change score indicates less pain. The SF-12 is a widely used preference-based utility measure of health derived from the SF-36.
Time Frame: baseline, 6 months, 12 months
Population: Sample size changes across cells due to attrition from baseline to 12 month interview.
Measure: Mean (Standard Deviation); unit: Changed mean z-score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed mean z-score
  Baseline to 6 months | -.16 (.75) | .11 (.86)
  6 months to 12 months: number analyzed (Participants) | 53 | 50
  6 months to 12 months | .19 (.91) | -.18 (.82)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change of z-scores; Test type: Superiority; p = .073, t-test, 2 sided
Statistical Analysis 2: Comparison: Health Navigation; Within-group mean z-score change from 6 months to 12-months (post-intervention) for the immediate treatment group only; Test type: Superiority; p = .066, t-test, 2 sided; Mean Difference (Net) = .19, Standard Deviation .91

2. Primary Outcome: Changed Health Screenings From Baseline to 6 Months and 12 Months
Description: Changed health screenings (e.g., pap smear, diabetes screening, blood pressure) from baseline to 6 months and 12 months for active intervention group and from 6 months to 12 months for waitlist control group. Clients select from a list of 8 possible routine screenings for ones they have completed in the last 6 months or since their last assessment. A higher change score indicates an increased rate of health screenings (which could reflect better care) and a lower score indicates fewer health screenings. Scores ranged from -6 to 7.
Time Frame: baseline, 6 months, 12 months
Population: There was differential attrition from baseline to 6 months and 6 months to 12 months.
Measure: Mean (Standard Deviation); unit: Changed count of health screenings
Groups:
- Health Navigation: 76 participants with SMI in the El Camino clinic, operated by Pacific Clinics, recruited to participate in a 12 month study of Bridge navigation. Randomly assigned to either waitlist control (6 month waitlist with treatment as usual) or immediate intervention with the Bridge. Participants in the immediate treatment group will complete three assessments (baseline, 6 months, and 12 months) and, after 6 months, one interview about their health, healthcare, and navigation experiences.
  Health Navigation: Experimental: Immediate peer health navigator intervention vs. waitlist control.
  The immediate peer health navigator intervention group will receive assistance for 6 months and then followed up with after an additional 6 months. Participants will receive training on how to self-manage their physical health and healthcare. The intervention is individualized and the number of contacts by the navigator will be determined by their need level.
- Waitlist Control: 75 participants with SMI in the El Camino clinic, operated by Pacific Clinics, were recruited to participate in a 12 month study. Randomly assigned to either waitlist control (6 month waitlist with treatment as usual then they will receive the intervention) or immediate intervention with the Bridge (n = 76). All participants completed 3 assessments (baseline, 6 month, 12 months) and one interview about their health, health care, and their experiences using health navigation after 12 months.
  Health Navigation: Experimental: Immediate peer health navigator intervention vs. waitlist control.
  The immediate peer health navigator intervention group received assistance for 6 months and then followed up with after an additional 6 months. Participants receive individual training on how to self-manage their physical health and healthcare. The waitlist control group completed a baseline assessment and then waited for 6 months before receiving the peer health naviga
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed count of health screenings
  Baseline to 6 months | .44 (2.35) | .45 (2.29)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | .17 (1.95) | .06 (2.37)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .983, t-test, 2 sided; Mean Difference (Final Values) = 0.022
Statistical Analysis 2: Comparison: Health Navigation; Within-group mean change from 6 months to 12-months (post-intervention) for the immediate treatment group only; Test type: Superiority; p = .533, t-test, 2 sided; Mean Difference (Net) = .17, Standard Deviation 1.95

3. Primary Outcome: Changed Number of Health Complaints From Baseline to 6 and 12 Months
Description: Changed number of Health Complaints from baseline to 6 and 12 months for the active intervention group and from 6 to 12 months by the waitlist control group. Participants will select yes/no whether they currently are experiencing any of 24 common health symptoms in the last 6 months. A count of the number of health complaints will be used in analyses. A negative change score would indicate a reduction in symptoms, which would indicate better health. Change scores ranged from -21 to 7.
Time Frame: baseline, 6 months, 12 months
Population: There was different attrition from baseline to 6 months and 6 months to 12 months.
Measure: Mean (Standard Deviation); unit: Changed mean of symptoms count
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed mean of symptoms count
  Baseline to 6 months | -1.07 (4.48) | -1.35 (4.81)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | .78 (3.60) | -.94 (4.13)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .731, t-test, 2 sided
Statistical Analysis 2: Comparison: Health Navigation; Within-group mean change from 6 months to 12-months (post-intervention) for the immediate treatment group only; Test type: Superiority; p = .211, t-test, 2 sided; Mean Difference (Final Values) = .29, Standard Deviation 1.67

4. Primary Outcome: Changed Scores on Health Care Efficacy Scale From Baseline to 6 Months and 12 Months
Description: Changed scores on The Health Care Efficacy Scale from baseline to 6 months and 12 months for the active intervention group and for the waitlist control group from 6 months to 12 months. This scale has been adapted from the Mental Health Confidence Scale, which was developed to measure the self-efficacy in individuals with a mental illness. This 14-item scale includes items on skills such as appointment making, pharmacy visits, establishing a medical home, and feeling that healthcare needs were heard and addressed. Participants will estimate the frequency of these experiences on a 3 point scale (1 = 'never' to 3 = '3 or more times'). A positive change score indicates improved health care self-efficacy.
Time Frame: baseline, 6 months, 12 months
Population: The sample size varied for comparisons overtime due to attrition.
Measure: Mean (Standard Deviation); unit: Change mean score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Change mean score
  Baseline to 6 months | .06 (.44) | .02 (.55)
  6 month to 12 months: number analyzed (Participants) | 48 | 47
  6 month to 12 months | .13 (.35) | -.02 (.36)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .244, t-test, 2 sided; Mean Difference (Net) = .04
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .016, t-test, 2 sided; Mean Difference (Net) = .13, Standard Deviation .35

5. Primary Outcome: Changed Score on Primary Care Provider Relationship From Baseline to 6 and 12 Months
Description: Changed ratings of a high-quality relationship with primary care providers from baseline to 6 and 12 months for active intervention group and from 6 months compared to 12 months for waitlist intervention group. Participants will be asked if they have a primary care provider (yes/no). Patients with a routine primary care provider will complete the Engagement with the Healthcare Provider Scale (as done with their navigator) regarding their relationship with their primary care provider. Mean scores range from 1 to 5 and the reported scores reflect the change in those scores from baseline to 6 months and 6 months to 12 months. A negative score indicates fewer issues with their healthcare provider over time in terms of units on a scale.
Time Frame: baseline, 6 months, 12 months
Population: The sample size varies across the timepoints due to attrition.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 44 | 46
Score on a scale
  Baseline to 6 months | -0.32 (.81) | .08 (.75)
  6 months to 12 months: number analyzed (Participants) | 42 | 37
  6 months to 12 months | .05 (.66) | -.17 (.69)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .019, t-test, 2 sided; Mean Difference (Net) = .40
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .609, t-test, 2 sided; Mean Difference (Net) = .05, Standard Deviation .66

6. Secondary Outcome: Changed Scores on Provider Level Stigma From Baseline in Comparison to 6 and 12 Months
Description: Changed ratings of provider stigma from baseline to 6 and 12 months for the immediate treatment group and from 6 months to 12 months for the waitlist control group. Provider-level stigma will be measured with a scale adapted from a provider level stigma scale in individuals with HIV/AIDS. This 7-item scale measures the degree to which clients experience stigma when they interact with health care providers, with items adapted to reflect SMI rather than HIV/AIDS. Participants rate their stigmatizing experiences with their provider on a 5-point scale (1= 'strongly disagree' to 5 = 'strongly agree'). Mean scores range from 1 to 5 with higher scores indicating agreement with experiences of stigma.
Time Frame: baseline, 6 months, 12 months
Population: The sample size varies across time points due to attrition.
Measure: Mean (Standard Deviation); unit: Mean change score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 44 | 46
Mean change score
  Baseline to 6 months | .06 (.62) | -.12 (.75)
  6 months to 12 months: number analyzed (Participants) | 44 | 38
  6 months to 12 months | -.06 (.59) | .13 (.60)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .203, t-test, 2 sided
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .480, t-test, 2 sided; Mean Difference (Net) = -.06, Standard Deviation .59

7. Secondary Outcome: Changed Scores of General Life Satisfaction From Baseline to 6 and 12 Months
Description: Changed scores of life satisfaction by the immediate treatment group from baseline to 6 and 12 months and from 6 months to 12 months for the waitlist control group. The Satisfaction with Life scale (SWL) is an 18-item Likert scale which measures participants' satisfaction with life in four domains: living situation, social relationship, work, and self and present life. It has shown good inter-item reliability (alpha = .88) and factorial validity in studies of the SMI. Mean scores range from 1 to 5, with higher scores indicating greater satisfaction with life. Change scores ranged from -1.42 to 1.59 with higher scores indicating an improvement over time in life satisfaction.
Time Frame: baseline, 6 months, 12 months
Population: The sample size varies across rows due to attrition over 12 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 58 | 59
Score on a scale
  Baseline to 6 months | .11 (.61) | .12 (.54)
  6 months to 12 months: number analyzed (Participants) | 51 | 43
  6 months to 12 months | .01 (.48) | .04 (.57)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .897, t-test, 2 sided; Mean Difference (Net) = .01
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .903, t-test, 2 sided; Mean Difference (Net) = .01, Standard Deviation .48

8. Secondary Outcome: Changed Scores on BASIS-24 From Baseline in Comparison to 6 and 12 Months
Description: Changed ratings of issues from baseline in comparison to 6 and 12 months assessments for immediate intervention group and from 6 months to 12 months for waitlist control group. The functional outcomes of the clients will be measured with the BASIS-24 (Behavior and Symptom Identification Scale). The 24 items of the BASIS-32 have been designed to assess a client's perception of difficulty due to psychiatric symptoms and problems in functional areas (daily living skills, work, and social) over the past week. Higher scores indicate greater difficulty. Scores range from 0 to 4. Change scores range from -2.18 to 1.58 with a positive score indicating an increase in difficulties.
Time Frame: baseline, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 60 | 60
Score on a scale | -.23 (.50) | -.15 (.62)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .433, t-test, 2 sided; Mean Difference (Net) = -.787
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .936, t-test, 2 sided; Mean Difference (Net) = .01, Standard Deviation .52

9. Secondary Outcome: Changed Unhealthy Habits From Baseline to 6 and 12 Months
Description: Using 1 item adapted from the National Leisure Time Survey, participants rated on a 7 point scale (0 = 'never' to 7 = 'daily') the frequency that participants exercise and scores were converted into z scores. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of more exercise. A negative change score indicates less exercise
Time Frame: baseline, 6 months, 12 months
Population: Exercise changed.
Measure: Mean (Standard Deviation); unit: Changed z-score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed z-score
  Baseline to 6 months | .18 (.95) | .04 (.79)
  6 months to 12 months: number analyzed (Participants) | 53 | 50
  6 months to 12 months | .07 (1.03) | -.16 (.89)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change in z-scores of diet; Test type: Superiority; p = .228, t-test, 2 sided
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .617, t-test, 2 sided; Mean Difference (Net) = .07, Standard Deviation 1.03

10. Secondary Outcome: Changed Scores of Internalized Stigma From Baseline to 6 and 12 Months
Description: Lower ratings of internalized stigma from baseline to 6 and 12 months for immediate intervention group and from 6 to 12 months for the waitlist control group. The 'Internalized Stigma of Mental Illness' scale (ISMI) will measure the internalized stigma of the clients along 5 dimensions of internalized stigma-alienation, stereotype endorsement, discrimination experience, social withdrawal and stigma resistance. Mean scores ranged from 1 to 4 with higher scores indicating a higher level of self-stigma. Change scores ranged from -.88 to 1.13, with negative change scores indicating a decrease in internalized stigma and a positive score indicating an increase in internalized stigma.
Time Frame: baseline, 6 months, 12 months
Population: The sample size changes due to attrition over time.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 60 | 61
Score on a scale
  Baseline to 6 months | .07 (.38) | .06 (.33)
  6 months to 12 months: number analyzed (Participants) | 53 | 48
  6 months to 12 months | .01 (.46) | .02 (.40)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .894, t-test, 2 sided; Mean Difference (Net) = .01
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .930, t-test, 2 sided; Mean Difference (Net) = .01, Standard Deviation .46

11. Secondary Outcome: ChangedPrescribed Medications From Baseline to 6 and 12 Months
Description: A decrease in medications is expected from baseline to 6 and 12 months for immediate treatment group and for the waitlist control group from 6 months to 12 months. Current medications are recorded for their name, dosage, frequency, timing, dates started, side effects noted, and reasons prescribed. A positive score indicates an increase in medications and a negative change score indicates a reduction in medications.
Time Frame: baseline, 6 months, 12 months
Population: The sample size changes due to attrition over the study period.
Measure: Mean (Standard Deviation); unit: changed count of medications
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
changed count of medications
  Baseline to 6 months | -.05 (1.16) | .10 (1.40)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | .24 (2.07) | -.04 (1.03)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .530, t-test, 2 sided; Mean Difference (Net) = .15
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .458, t-test, 2 sided; Mean Difference (Net) = -.13, Standard Deviation 1.27

12. Secondary Outcome: Changed Number of Health Diagnoses From Baseline to 6 and 12 Months
Description: Changed rates of identification of previously undetected chronic health conditions, decreased number of other disorders from baseline to 6 and 12 months in active intervention group and from 6 to 12 months in the waitlist control group. Changes in the number of diagnoses ranged from -3 to 5. Positive changes indicate an increased in diagnosed conditions and negative scores indicate a reduction in diagnoses.
Time Frame: baseline, 6 months, 12 months
Population: The sample changes over time due to attrition.
Measure: Mean (Standard Deviation); unit: Changed count of conditions
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed count of conditions
  Baseline to 6 months | .23 (.69) | -.08 (.91)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | .02 (1.00) | -.34 (1.26)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .036, t-test, 2 sided; Mean Difference (Net) = .31
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .892, t-test, 2 sided; Mean Difference (Net) = .02, Standard Deviation 1.00

13. Secondary Outcome: Changed Euroqual Health Score From Baseline to 6 and 12 Months
Description: Changed rating of Euroqual health score from baseline to 6 and 12 months by active intervention group and from 6 months to 12 months for the waitlist control group. Participants rate their health from highest possible to worst possible from 100 to 0. Change scores ranged from -90 to 100. Positive scores indicate better health and negative scores indicate worsening health.
Time Frame: baseline, 6 months, and 12 months
Population: The sample size changed over time due to attrition.
Measure: Mean (Standard Deviation); unit: Changed mean score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Changed mean score
  Baseline to 6 months | 3.70 (21.78) | 3.29 (30.55)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | -6.43 (24.34) | 7.12 (20.90)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .931, t-test, 2 sided; Mean Difference (Net) = .41
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .058, t-test, 2 sided; Mean Difference (Net) = -6.43, Standard Deviation 24.34

14. Secondary Outcome: Changed Euroqual Satisfaction With Provider Score From Baseline to 6 and 12 Months
Description: Changed rating of Euroqual satisfaction with provider score from baseline to 6 and 12 months by active intervention group and from 6 months to 12 months for the waitlist control group. Participants rate their satisfaction from highest possible to worst possible from 100 to 0. Change scores ranged from -90 to 79. Positive scores indicate improved satisfaction and negative scores indicate declines in satisfaction.
Time Frame: baseline, 6 months, and 12 months
Population: The sample size differs over time due to attrition.
Measure: Mean (Standard Deviation); unit: Mean change score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 48 | 51
Mean change score
  Baseline to 6 months: number analyzed (Participants) | 47 | 51
  Baseline to 6 months | 6.32 (28.76) | 2.71 (34.43)
  6 months to 12 months: number analyzed (Participants) | 48 | 50
  6 months to 12 months | -1.06 (33.89) | 7.12 (20.9)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Test type: Superiority; p = .576, t-test, 2 sided; Mean Difference (Net) = .40
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .829, t-test, 2 sided; Mean Difference (Net) = -1.06, Standard Deviation 33.89

15. Secondary Outcome: Changed Substance Use From Baseline to 6 and 12 Months
Description: Changed substance use from baseline to 6 and 12 months for the immediate treatment group and for the waitlist control group from 6 months to 12 months (e.g., alcohol, nicotine, cocaine, marijuana, prescription drugs). Scores ranged from 0 to 9, with a higher number indicating a greater variety of substances used. A negative score indicates a reduced variety of substances used and a positive score indicates an increase in the variety of substances used (range from -2 to 2 for change scores).
Time Frame: baseline, 6 months, 12 month
Population: Sample changed over time due to attrition
Measure: Mean (Standard Deviation); unit: Count of substances
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Count of substances
  Baseline to 6 months | -.08 (.81) | -.13 (.84)
  6 months to 12 months: number analyzed (Participants) | 53 | 50
  6 months to 12 months | .04 (.55) | -.11 (.32)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .792, t-test, 2 sided
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .622, t-test, 2 sided; Mean Difference (Net) = .04, Standard Deviation .55

16. Secondary Outcome: Changed Score on Self Management Motivation
Description: Changed score on Self Management Motivation scale from baseline to 6 months and 12 months in active intervention group and changed score from 6 months to 12 months in the waitlist control group. 9 item measure written for this study. Participants rate how important and how confident they are about managing their health (1 = not at all confident to 10 = very confident). Changes in confidence ranged from -4.44 to 4.00. Positive scores indicate an increased confidence and negative scores indicate a decrease in confidence.
Time Frame: baseline, month 6, month 12
Population: The sample sizes differ over time due to attrition.
Measure: Mean (Standard Deviation); unit: Mean change score
Arm/Group | Health Navigation | Waitlist Control
Number analyzed (Participants) | 61 | 62
Mean change score
  Baseline to 6 months | .33 (1.65) | -.28 (.78)
  6 months to 12 months: number analyzed (Participants) | 54 | 50
  6 months to 12 months | .29 (1.67) | .57 (1.81)
Statistical Analysis 1: Comparison: Health Navigation vs Waitlist Control; Baseline to 6 months between-group comparisons of the mean change; Test type: Superiority; p = .049, t-test, 2 sided; Mean Difference (Net) = 1.986
Statistical Analysis 2: Comparison: Health Navigation; Test type: Superiority; p = .211, t-test, 2 sided; Mean Difference (Net) = .29, Standard Deviation 1.67

ADVERSE EVENTS:
Groups:
- Health Navigation: 76 participants with SMI in the El Camino clinic, operated by Pacific Clinics, recruited to participate in a 12-month study of Bridge navigation. Randomly assigned to either waitlist control (6 month waitlist with treatment as usual) or immediate intervention with the Bridge. All participants complete 3 assessments (baseline, 6 months, and 12 months) and, after 6 months, one interview about their health, healthcare, and navigation experiences.
  Health Navigation: Experimental: Immediate peer health navigator intervention vs. waitlist control.
  The immediate peer health navigator intervention group will receive assistance for 6 months and then followed up with after an additional 6 months. Participants will receive training on how to self-manage their physical health and healthcare. The intervention is individualized and the number of contacts by the navigator will be determined by their need level.
- Waitlist Control: 75 participants with SMI in the El Camino clinic, operated by Pacific Clinics, will be recruited to participate in a 12 month study of Bridge navigation. Randomly assigned to a waitlist control condition (6-month waitlist with treatment as usual then they receive the intervention) and completed 3 assessments (baseline, 6 month, 12 months) and one interview about their health, health care, and their experiences using health navigation after 12 months.
Arm/Group | Health Navigation | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 1/76 | 2/75
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

LIMITATIONS AND CAVEATS:
Limited to a single mental health agency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No